CLINICAL TRIAL: NCT02935023
Title: Carbon Ion Radiotherapy in Treating Patients Undergoing Systemic Therapy for Oligo-metastatic Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Shen Fu, Director,department of radiation oncology, Shanghai Proton and Heavy Ion Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-PCa2016-01
Record Dates: First submitted 2016-10-11; First posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Metastatic Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CIRT with systemic therapy arm (Experimental): Carbon ion radiotherapy combined with systemic therapy
  Interventions: Radiation: CIRT with systemic therapy arm

INTERVENTIONS:
Radiation: CIRT with systemic therapy arm — carbon ion radiotherapy to the prostate(59.2GyE/16Fx to prostate and seminal vesicle) Systemic therapy:Hormonal therapy (LHRH agonist and/or antiandrogens) or chemotherapy

SUMMARY:
The goal of this clinical study is to determine impact of carbon ion radiotherapy (CIRT) treatment in combination with systemic therapy for oligo-metastatic prostate cancer. The primary objective: to determine disease biochemical progression-free survival in man with oligo-metastatic (M1a/b) prostate cancer undergoing systemic therapy with definitive radiotherapy of the primary tumor. The secondary objective: to determine local control, overall survival and quality of life in men with oligo-metastatic prostate cancer undergoing carbon ion radiotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed adenocarcinoma of the prostate
2. Age ≥ 20 and < 80 years of age
3. ECOG PS 0 or 1
4. Life-expectancy ≥1 year
5. Stage T1-4,N0-1,M1a/b disease on imaging, with a combined maximum of 3 synchronous lesions.
6. Ability to understand and willingness to sign informed consent

Exclusion Criteria:

1. No pathologically confirmed adenocarcinoma of the prostate
2. visceral metastasis
3. Previous pelvic radiotherapy or prostatectomy
4. Severe systemic disorders

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Time to PSA relapse | From the start of systemic therapy, a median of 2 years

SECONDARY OUTCOMES:
progression free survival | From the start of systemic therapy, a median of 2 years
Overall survival | From the start of systemic therapy, a median of 2 years
Quality of life | From the start of carbon ion radiotherapy, a median of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shen Fu, PhD.MD., Study Director — Shanghai Proton and Heavy Ion Center
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No